CLINICAL TRIAL: NCT02647086
Title: An Open-Label, Drug-Drug Interaction Study to Examine the Effects of Dupilumab on the Pharmacokinetics of Selected Cytochrome P450 Substrates in Adult Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Open Label, Drug-Drug Interaction (DDI) Study of Dupilumab (REGN668/SAR231893) in Patients With Moderate to Severe Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R668-AD-1433
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Atopic Dermatitis
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — dupilumab; Midazolam; Omeprazole; Warfarin; Caffeine; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period 1 (Experimental): Patients will receive selected Cytochrome P450 substrates (Midazolam, Omeprazole, Warfarin, Caffeine, Metoprololin) in period 1 (day 1)
  Interventions: Drug: Midazolam; Drug: Omeprazole; Drug: Warfarin; Drug: Caffeine; Drug: Metoprolol
- Period 2 (Experimental): Patients will receive dupilumab starting in Period 2 (day 8) and continue weekly through day 50; Patients will receive selected Cytochrome P450 substrates (Midazolam, Omeprazole, Warfarin, Caffeine, Metoprolol) in period 2 (at day 36).
  Interventions: Drug: Dupilumab; Drug: Midazolam; Drug: Omeprazole; Drug: Warfarin; Drug: Caffeine; Drug: Metoprolol

INTERVENTIONS:
Drug: Dupilumab
  Other Names: REGN668/SAR231893
  Arms: Period 2
Drug: Midazolam — Cytochrome P450 substrate
Drug: Omeprazole — Cytochrome P450 substrate
Drug: Warfarin — Cytochrome P450 substrate
Drug: Caffeine — Cytochrome P450 substrate
Drug: Metoprolol — Cytochrome P450 substrate

SUMMARY:
This is an open-label, single-sequence DDI study designed to examine the effects of dupilumab on the pharmacokinetics of selected cytochrome P450 substrates in adult patients with moderate to severe AD.

The study consists of a screening period (day -35 to -2), study period 1 (day -1 to 7), study period 2 (day 8 to 50), and a follow-up period (day 51 to 135 [end of study]).

Following completion of study period 2 (Day 50), patients will be given the option to enroll into the Open-Label Extension (OLE) study R668-AD-1225. Patients who decline will be followed for the next 12 weeks (Day 135).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient, aged 18 years or older
2. Diagnosis of Chronic AD, defined as diagnosis of AD for at least 3 years before the screening visit
3. Eczema Area Severity Index (EASI) score ≥16 at the screening and baseline visits
4. Investigator's Global Assessment (IGA) score ≥3 (on the 0 to 4 IGA scale) at the screening and baseline visits
5. ≥10% Body Surface Area (BSA) of AD involvement at the screening and baseline visits
6. Patients with documented recent history (within 6 months before the screening visit) of inadequate response to outpatient treatment with topical medications, or for whom topical treatments are otherwise medically inadvisable (eg, because of important side effects or safety risks)
7. Provide signed informed consent

Exclusion Criteria:

1. Prior participation in a dupilumab clinical trial
2. The use of any of the following treatments within 4 weeks before the baseline visit:

   * Systemic corticosteroids
   * Immunosuppressive/immunomodulating drugs
   * Phototherapy for AD
3. Administration, within 14 days before baseline or within a period of 5 times the elimination half-life of the medication before baseline, whichever is longer, of any medication that is a known inducer or inhibitor of either one or more of the following CYP enzymes: CYP3A, CYP2C19, CYP2C9, CYD2D6, and CYP1A2. Patients who are on any of these medications at the time of screening and cannot be safely taken off these medications will be excluded from the study.
4. Any contraindication to one or more of the following drugs, according to the applicable labeling:

   * Midazolam
   * Omeprazole
   * Warfarin
   * Caffeine
   * Metoprolol
5. Consumption of any 1 or more of the following food items and/ or beverages within 1 week prior to baseline:

   * Grapefruit or grapefruit juice, apple or apple juice, orange or orange juice, lemons or lemon juice, limes or lime juice
   * Vegetables from the mustard green family (eg, broccoli)
   * Charbroiled meats
   * Caffeinated beverages, foods or drugs containing caffeine Patients who are not willing to abstain from the consumption of these food items and/or beverages for certain periods during the study will also be excluded
6. History of excessive consumption of beverages containing caffeine (more than 4 cups or glasses per day). Patients who are not willing to abstain from the consumption of caffeine during certain periods of the study will also be excluded
7. History or presence of alcohol or drug abuse within last 2 years
8. History of smoking within last 2 years
9. Poor metabolizers for CYP2C9, CYP2C19, or CYP2D6 based on genotyping
10. Presence of any one or more of the following lab abnormalities at screening:

    * Platelet count ≤100 x 10^3/µL
    * Neutrophils ≤1 x 10^3/µL
    * Creatinine phosphokinase (CPK) >10 x upper limit of normal (ULN)
    * International normalized ratio (INR) ≥2
11. Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiprotozoals, or antifungals within 2 weeks before the screening visit, or superficial skin infections within 1 week before the screening visit
12. Known or suspected immunodeficiency, including history of invasive opportunistic infections (eg, tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution, or otherwise recurrent infections of abnormal frequency or prolonged duration suggesting an immune compromised status, as judged by the investigator
13. History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening
14. Positive with hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody (Hep C Ab) at the screening visit. NOTE: Patients who are HBsAg negative and HBsAb positive are considered immune after a natural infection has cleared or they have been vaccinated against hepatitis B. Therefore, they are acceptable for the study.
15. History of malignancy within 5 years before the baseline visit, except completely treated in situ carcinoma of the cervix, and completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin
16. History of clinical endoparasitosis (ie, helminth infection) within 12 months before the baseline visit, or high risk of helminth infection, such as residence within or recent travel (within 12 months before the baseline visit) to areas endemic for endoparasitoses, where the circumstances are consistent with parasite exposure (eg, extended stay, rural or slum areas, lack of running water, consumption of uncooked, undercooked, or otherwise potentially contaminated food, close contact with carriers and vectors, etc), unless subsequent medical assessments (eg, stool exam, blood tests, etc) have ruled out the possibility of parasite infection/infestation
17. Female patients who are pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study
18. Women who are using any form of hormonal contraceptives (eg, oral, injectables, implants, patches, rings, hormone-impregnated intrauterine devices [IUDs]) for birth control
19. Women unwilling to use adequate birth control, if of reproductive potential and sexually active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Ratio of Area Under Curve last (AUClast) and maximum concentration (Cmax) for Cytochrome P450 substrates from pre-dupilumab administration at baseline (period 1, day 1) | At Baseline (day 1)
Ratio of AUClast and Cmax for CYP substrates 4 weeks after initiating a weekly regimen of dupilumab (period 2, day 36) | At day 36

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) from day of first administration of dupilumab to end of study (day 50 for patients who enroll in the OLE study; day 134 for patients who decline participation in the OLE). | Baseline up to day 134

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (5):
- United States (5):
  - Regeneron Study Site, Little Rock, Arkansas
  - Regeneron Study Site, Centennial, Colorado
  - Regeneron Study Site, Minneapolis, Minnesota
  - Regeneron Study Site, Berlin, New Jersey
  - Regeneron Study Site, Raleigh, North Carolina

REFERENCES:
- [Derived] Davis JD, Bansal A, Hassman D, Akinlade B, Li M, Li Z, Swanson B, Hamilton JD, DiCioccio AT. Evaluation of Potential Disease-Mediated Drug-Drug Interaction in Patients With Moderate-to-Severe Atopic Dermatitis Receiving Dupilumab. Clin Pharmacol Ther. 2018 Dec;104(6):1146-1154. doi: 10.1002/cpt.1058. Epub 2018 Apr 2. PMID 29498038